CLINICAL TRIAL: NCT07371390
Title: Minimal Sedation During Total Knee Arthroplasty: A Prospective Randomized Control Trial
Brief Title: Minimal Sedation During Knee Replacement Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Professor of Orthopedics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-010602
Record Dates: First submitted 2025-12-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Arthroplasty
Keywords: Spinal Anesthesia; Minimal Sedation; Total Knee Arthroplasty; Knee Replacement; Audiovisual Distraction; Localized Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No active noise cancelling headset (No Intervention): This arm will serve as the control group for this randomized trial. Patients in this arm will receive normal standard of care anesthesia during their total knee arthroplasty.
- Active Noise Cancelling Headset (Experimental): This arm will provide patients with an active noise cancelling headset system that they may use to select music or a movie for audiovisual distraction during the surgery.
  Interventions: Device: Active Noise Cancelling Headset System

INTERVENTIONS:
Device: Active Noise Cancelling Headset System — The ANC Headset will allow patients to select music or a movie for audiovisual distraction during their surgery. This can be used when patients are not receiving general anesthesia (full sedation) for their surgery.
  Arms: Active Noise Cancelling Headset

SUMMARY:
This study will test the use of active noise cancelling headphones with music or a movie during knee replacement surgery. Feedback from the surgical team and from patients regarding the headset system will be gathered to see if using it can reduce the amount of sedation needed during knee replacement procedures that use localized anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Primary Total Knee Arthroplasty
* Indicated for Spinal Anesthesia
* 18+ years old
* Participant can independently provide informed consent

Exclusion Criteria:

* Unicompartmental Knee Arthroplasty
* Revision Knee Arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean Richmond Agitation-Sedation Scale(RASS) Score | 30 minutes intraoperatively
  Richmond Agitation-Sedation Scale (RASS) measures the amount of sedation necessary for a patient at different levels of discomfort or agitation during local anesthesia surgeries.
Protocol Completion | Intraoperatively
  This will measure the volume of patients that were unable to complete their procedure using spinal anesthesia and due to discomfort or agitation required deep sedation to continue to surgery.
Mean Propofol Infusion Rate | Intraoperatively
  Mean rate of propofol infusion necessary to achieve sedation targets during the procedure. Unit: mcg/kg/min

SECONDARY OUTCOMES:
Patient Satisfaction | Within 48 hours post-operatively
  Patients will complete a satisfaction questionnaire post-operatively to determine their level of comfort with the sedation protocol they received during surgery.
Surgeon Satisfaction | Within 48 hours post-operatively
  Surgeons will be asked if they experienced interruptions or difficulty completing the procedure due to the sedation protocol administered to the patient.
Anesthetist Satisfaction | Within 48 hours post-operatively
  Anesthesia staff will receive a questionnaire regarding satisfaction with efficacy of the sedation protocol administered during the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Abdel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided, as publication plan has not been finalized at this time.